CLINICAL TRIAL: NCT03470623
Title: Randomized, Prospective Comparison of Bioabsorbable and Steel Screw for the Treatment of Hallux Valgus With Chevron Osteotomy
Brief Title: Comparison of Bioabsorbable and Steel Screw for the Treatment of Hallux Valgus With Chevron Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00123456
Record Dates: First submitted 2018-03-10; First posted 2018-03-20 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Hallux Valgus
Keywords: hallux valgus; chevron osteotomy; bioabsorbable screw; steel screw
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bioabsorbable screws (Experimental): hallux valgus treated with chevron osteotomy using bioabsorbable screws
  Interventions: Device: bioabsorbable screws
- steel screws (Experimental): hallux valgus treated with chevron osteotomy using steel screws
  Interventions: Device: steel screws

INTERVENTIONS:
Device: bioabsorbable screws — Hallux valgus are treated with a distal chevron osteotomy of first metatarsal and fixed using the bioabsorbable screw
  Arms: bioabsorbable screws
Device: steel screws — Hallux valgus are treated with a distal chevron osteotomy of first metatarsal and fixed using the steel screw
  Arms: steel screws

SUMMARY:
Hallux valgus is the most common deformity of forefoot and the patients would suffer pain and disable of walking and wearing normal shoes. Chevron osteotomy of the first metatarsal is widely used for the treatment of mild or medium hallux valgus. It is a "V" sharp osteotomy that can decrease the intermetatarsal degree of first-second metatarsal by pushing the distal side of osteotomy laterally.A 2.5mm or 3.0mm steel cannulated screw is usually used for the fixation of the osteotomy side to provide stability.However,there are some shortcomings of steel screws such as rejection of internal fixation or the financial cost of the second surgery of fixation taken-out. To obviate these shortcomings of steel screws, bioabsorbable screw fixation may be an alternative method for chevron osteotomy.

This trial is a randomized, prospective, controlled, parallel experimental design, to compare the clinical and radiographic outcomes of bioabsorbable screw versus steel screw for the treatment of hallux valgus with chevron osteotomy. The patients will be randomized to two groups, one treated with bioabsorbable screws while the other treated with steel screws.Data collection for the outcomes measures will occur pre-op,immediate post-op and then 6 weeks, 12 weeks, and at 1 years post operation.

The clinical outcomes measure are the VAS (visual analogue scale) score and AOFAS (American orthopedic foot and ankle society) forefoot score.The radiographic outcomes measures are the IMA (intermetatarsal angle) and the HVA (hallux valgus angle)

ELIGIBILITY:
Inclusion Criteria:

1. hallux valgus treated with distal chevron osteotomy
2. age between 18-70

Exclusion Criteria:

1. hallux valgus treated with other procedure (scarf,ludloff,lapidus,etc)
2. age <18 or age >70
3. rheumatoid
4. osteoporosis -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
American orthopedic foot and ankle society forefoot score change | pre-op,6 weeks,12 weeks and 1 year after operation
  American orthopedic foot and ankle society forefoot score was consist of "pain","ability of walking" and "alignment".The minimum score is 0 and the maximum score is 100, "0"means worst while "100" means best of the outcome. It was used as a standard evaluation method of hallux valgus.

SECONDARY OUTCOMES:
Radiographic outcomes parameters | pre-op,6 weeks,12 weeks and 1 year after operation
  IMA (intermetatarsal angle ),HVA (hallux valgus angle) measured in weight-bearing anteroposterior of foot
VAS score | pre-op,6 weeks,12 weeks and 1 year after operation
  Visual Analogue Scale,a widely used score about pain. It present different level of pain by using the number 0-10. 0 present no pain while 10 present worst pain

IPD SHARING:
Plan to Share IPD: Yes